CLINICAL TRIAL: NCT07226505
Title: A Randomized Trial Analyzing the Effects of Core Strengthening Exercises in Physical Therapy for Treating Temporomandibular Joint Dysfunction
Brief Title: Effects of Core Strengthening Exercises for Treating TMD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Loyola University (Other)
Collaborators: Loyola University Chicago (Other)
Responsible Party: Principal Investigator, Margaret Miller, MD, Loyola University Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 219911
Record Dates: First submitted 2025-10-30; First posted 2025-11-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-10

CONDITIONS: Temporomandibular Joint Dysfunction; TMD; TMJ Internal Derangement; Myofascial Pain
Keywords: Core strengthening; physical therapy; RCT
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Who Masked: Participant
Masking Description: Single-blinded (evaluating PT blinded)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Core Strengthening + Standard TMD Physical Therapy (Experimental): Participants in this group will receive the Shirley Sahrmann core strengthening protocol, which involves progressive levels of dynamic movements designed to maintain a neutral spine and activate deep core muscles. Exercises begin in hook-lying or supine positions, with gradual progression through five levels, and may include upper extremity movements once core control is achieved. In addition, participants will follow a structured home exercise program with daily exercises (approximately 20 minutes), supported with printed instructions and video demonstrations through the MedBridge platform.
  Interventions: Behavioral: Experimental: Group 1: Core Strengthening; Behavioral: Group 2: Standard TMD PT
- Group 2: Standard TMD Physical Therapy (Active Comparator): Participants in this group will receive standard physical therapy for TMD, including:
  Therapeutic exercises (e.g., Rocabado 6x6) for jaw mobility and posture.
  Manual therapy to restore normal TMJ and cervical spine joint mechanics.
  Soft tissue mobilization targeting masticatory and cervical muscles as clinically indicated.
  Education on jaw rest position, diet/chewing modifications, and avoidance of parafunctional habits.
  Neuromuscular re-education to improve TMJ opening mechanics, including deep neck flexor activation and mirror training.
  Interventions: Behavioral: Group 2: Standard TMD PT

INTERVENTIONS:
Behavioral: Experimental: Group 1: Core Strengthening — Participants perform Shirley Sahrmann core exercises (5 progressive levels maintaining neutral spine and deep core activation), possibly adding upper extremity movements. Standard TMD PT includes jaw exercises, manual therapy, soft tissue mobilization, neuromuscular re-education, and patient education. A home exercise program (~20 min/day) is provided with printed and video instructions.
  Other Names: Shirley Sahrmann Core Stability Protocol
  Arms: Group 1: Core Strengthening + Standard TMD Physical Therapy
Behavioral: Group 2: Standard TMD PT — Participants receive standard TMD PT including jaw exercises (Rocabado 6x6), manual therapy for TMJ and cervical spine, soft tissue mobilization, neuromuscular re-education to improve jaw mechanics, and education on jaw positioning, diet/chewing modifications, and parafunctional habits. A home exercise program is provided as part of treatment.
  Other Names: Rocabado 6x6 Exercises

SUMMARY:
Temporomandibular disorders (TMD) are commonly managed with non-invasive interventions such as manual therapy, therapeutic exercise, relaxation techniques, and patient education. Core strengthening (also known as abdominal strengthening) is a fundamental element of physical therapy that engages deep and superficial trunk musculature to enhance postural control and functional performance. Protocols such as the Shirley Sahrmann progression have demonstrated increased activation of key core stabilizing muscles. Emerging evidence suggests a potential relationship between core stability training and reductions in TMD-related pain, though improvements in functional outcomes remain inconclusive. Biomechanical links between the pelvic floor, spine, and temporomandibular joint further support the rationale for core-focused interventions. Nevertheless, few studies have isolated the effects of core strengthening on TMD symptomatology. This study seeks to determine whether the integration of core stability exercises into TMD management can reduce pain, improve function, and enhance quality of life.

DETAILED DESCRIPTION:
This single-blinded randomized controlled trial will evaluate the effects of core strengthening exercises in addition to standard physical therapy for patients with Temporomandibular Joint Dysfunction (TMD). The study aims to determine whether integrating core stability exercises can reduce TMD-related pain, improve function, and enhance quality of life compared to standard physical therapy alone.

A total of 50 participants, aged 18-70, who have a primary complaint of TMD within the last 30 days and are willing to complete at least six physical therapy visits over a three-month period will be enrolled. Participants must speak English or have access to a verified interpreter and be able to safely participate in exercise.

Participants will be randomly assigned to one of two groups:

Group 1: Core strengthening exercises (Shirley Sahrmann progression) combined with standard TMD physical therapy, including therapeutic exercises, manual interventions, soft tissue mobilization, neuromuscular re-education, and education. Home exercise programs will support adherence.

Group 2: Standard TMD physical therapy alone, including the same therapeutic exercises, manual interventions, soft tissue mobilization, neuromuscular re-education, and education.

Key exclusion criteria include recent TMJ or spinal surgery, recent head/neck trauma or neurologic symptoms, pregnancy, concurrent physical therapy for other movement disorders, low back or pelvic health dysfunction in the past three months, use of dentures, or current chemotherapy/radiation involving the head, neck, pelvis, spine, or hip.

Participants will undergo initial evaluation, intervention sessions, and post-treatment assessment by blinded evaluating therapists to measure pain, function, and core strength outcomes. Safety will be continuously monitored throughout the study.

ELIGIBILITY:
Who Can Participate (Inclusion Criteria):

Adults between 18 and 70 years old.

Have had jaw pain or problems with the jaw joint (TMD) in the last 30 days.

Able and willing to attend at least six physical therapy sessions over three months.

Speak English or have access to a qualified interpreter.

Able to safely do physical exercises.

Who Cannot Participate (Exclusion Criteria):

Recently had surgery on the jaw, teeth, or spine (within the last 3 months).

Recently had head or neck injuries or certain neurological problems (such as dizziness, double vision, trouble swallowing, or sudden falls).

Are pregnant or become pregnant during the study.

Currently doing physical therapy for other movement problems that could affect the study.

Have had lower back or pelvic health issues in the last 3 months.

Currently receiving chemotherapy or radiation for cancer in the head, neck, pelvis, spine, or hip.

Wear dentures or cannot safely perform exercises.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
TMD Pain (e.g., Visual Analog Scale/Numeric Pain Rating) | Baseline and post-intervention (6 PT sessions), assessed up to 6 weeks

SECONDARY OUTCOMES:
Neck Disability Index (NDI) | Baseline and post-intervention (6 PT sessions), assessed up to 6 weeks
  This measure evaluates how neck pain affects a person's ability to perform everyday activities. It uses the Neck Disability Index (NDI), a questionnaire scored from 0% to 100%, where 0% means no disability and 100% represents complete disability in daily life.
Compliance with Home Exercise Program (HEP) | Throughout the 6-week intervention period (daily tracking, summarized at post-intervention)
  Assessed via participant-completed exercise diaries, tracking adherence to prescribed daily exercises.
Functional Measures from TMJ Scale | Baseline and post-intervention (6 PT sessions), assessed up to 6 weeks
  This measure objectively evaluates jaw movement and functional performance, including mobility, deviation, and deflection. It uses the Temporomandibular Disorder (TMD) Dysfunction Scale, which consists of 10 questions scored from 0 to 4. The total score is converted to a percentage, where higher percentages reflect greater levels of dysfunction or disability.

CONTACTS AND LOCATIONS:
Locations (1):
- Loyola University Medical Center, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No